CLINICAL TRIAL: NCT02224248
Title: The Effect of Including Fitness Testing in Preventive Health Checks on Cardiorespiratory Fitness and Motivation to Change Physical Activity Behaviour
Brief Title: Effect of Including Fitness Testing in Preventive Health Checks on Cardiorespiratory Fitness and Motivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Randers Municipality, Denmark (Other); Central Denmark Region (Other); TRYG Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1-15-1-72-13-09
Record Dates: First submitted 2014-08-08; First posted 2014-08-25 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2015-12

CONDITIONS: Cardiorespiratory Fitness; Physical Activity; Health Behavior; Motivation; Intention
Keywords: cardiorespiratory fitness; exercise tolerance; exercise test; health behavior; motor activity; motivation; intention; self-rated health
MeSH Terms: conditions — Motor Activity; Health Behavior | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Health checks with fitness testing (Experimental)
  Interventions: Behavioral: Health checks with fitness testing
- Health checks without fitness testing (Active Comparator)
  Interventions: Behavioral: Health checks without fitness testing

INTERVENTIONS:
Behavioral: Health checks with fitness testing — Fitness testing as part of a preventive health check compose the intervention in this trial. Thus, the intervention group will receive preventive health checks with fitness testing.
  Arms: Health checks with fitness testing
Behavioral: Health checks without fitness testing — The active comparator will not receive fitness testing as part of the preventive health checks. With the exception of fitness testing, the preventive health checks in the active comparator group and the intervention group are identical.
  Arms: Health checks without fitness testing

SUMMARY:
The purpose of this study is to investigate if including fitness testing in preventive health checks increase cardiorespiratory fitness and motivation to change physical activity behavior compared with preventive health checks without fitness testing.

DETAILED DESCRIPTION:
BACKGROUND

Changing unhealthy lifestyle improves health and reduces morbidity. Motivation is a key component in initiation and maintenance of lifestyle changes. Identifying and motivating individuals with unhealthy lifestyle to change behaviour may be achieved through preventive health checks as already implemented in some countries. However, knowledge about the impact of individual components included in preventive health checks is lacking. Consequently, the most effective composition of preventive health checks remains unknown.

In a Danish municipality, the Check your Health Prevention Program (CHPP) was recently initiated, offering preventive health checks to all 30 to 49 year-old citizens. This program provides the unique opportunity to evaluate single components of a preventive health check in a real-life setting. Only a few previous studies have included cardiorespiratory fitness (fitness) testing in a preventive health check. Fitness is associated with multiple health benefits such as improved cardio-metabolic profile and reduced risk of cancer, diabetes, and depression.

The investigators aim to investigate the effect of including fitness testing in preventive health checks on fitness level, motivation for changing physical activity behaviour, physical inactivity prevalence and self-rated health. The investigators hypothesize that fitness testing as part of preventive health checks compared to preventive health checks without fitness testing 1) increases fitness level assessed after one year and the percentage of participants increasing motivation to change physical activity behaviour assessed after two weeks, and 2) reduces physical inactivity prevalence and improves self-rated health scores during the one-year study period.

METHODS

Nested-design

The present trial is embedded in the above mentioned health promotion program, CHPP, which is conducted during the years 2012 to 2017. In the CHPP, all citizens living in the municipality of Randers aged 30-49 years per 1st of January 2012 (n = 26,216) were identified in the Danish Civil Registration System.The identified population was randomized into five equal groups, one for each year of the CHPP. Invitations are dispatched continuously by mail and include information about the CHPP and a prefixed appointment for a health check. Health checks and health behavioural courses will take place at Randers Health Centre and health consultations at the citizen´s general practitioner.

The health check

Besides the addition of fitness testing in the intervention group, the preventive health checks will include assessments of the following: body weight and height, waist circumference, blood pressure, lipid profile (total cholesterol, LDL, HDL, and triglycerides), HbA1c and lung function. Moreover, a baseline questionnaire regarding physical activity level, motivation for changing physical activity behaviour, self-rated health, smoking, and alcohol will be answered in connection with the health check. At the end of the health check, the results are presented in a personalized health profile leaflet, which includes recommendations for follow-up according to the risk-profile. The baseline questionnaire and the subsequent follow-up procedures are identical in the two study groups.

Standardization and education

The health check will be conducted by health professionals who have been trained in all measurement procedures as well as in risk communication to ensure standardization and quality. Execution of the health check is further standardized by a written protocol and adherence to the protocol is checked continuously. Furthermore, a process evaluation will be conducted.

Outcome assessment

Cardiorespiratory fitness will be assessed by submaximal cycle ergometer testing. Motivation for changing physical activity behavior will be assessed using the Transtheoretical Model´s Stages of Change, and secondary outcomes using a modified version of the questions developed by Saltin and Grimby and the Short-Form 12, Health Survey, version 2.

Follow up

All participants will receive a questionnaire regarding motivation for changing physical activity behaviour two weeks after the health check and will be invited for fitness testing after one year.

Randomization and blinding

Randomization is handled by a data-manager with no scientific involvement. The eligible population for this trial was defined by the CHPP randomization. Citizens randomized for the third out of five years of the CHPP will be further randomized by household to either intervention or control in the present trial. The intervention, the outcomes, group assignment, and the future outcome assessments in this trial are unrevealed in the invitation for the CHPP. The health behavioural courses and the health consultations will be carried out un-blinded due to the real-life setting. At the one-year follow-up, the personnel assessing the outcomes will be independent and blinded to group allocation.

Sample size

An estimated sample size of 1,500 participants allows for a categorical analysis of fitness level and is calculated on the basis of the following assumptions: 1:1 randomization, false positive error rate of 0.05, power of 0.8, intracluster correlation coefficient of 0.05 and categorical analysis with a power to detect a difference of 10% in the prevalence of very low fitness between the study groups. The investigators determined this 10% difference to be clinically meaningful based on expert opinions and criteria employed in other research. The intracluster correlation coefficient was included to reflect a possible clustering effect of the general practitioners (n = 46), which is seldom greater than 0.05 in primary care settings. The estimated sample size accounts for a 30% loss to follow-up.

Statistics

Statistical analysis will be performed using STATA 12.0 software. Continuous variables are presented as mean ±standard deviation and categorical variables as absolute numbers and relative (%) frequencies. In the comparative analyses Student´s t-test will be used, when comparing means or changes in means of continuous variables and Chi2-test or Fisher's exact t-test, when comparing proportions for categorical variables. Analyses will be adjusted for baseline physical activity. Stratified analyses will be performed on sex and age groups and analysis of motivation will only be performed on the subgroup comprising precontemplaters, contemplaters, and preparators at baseline. All analyses will follow the intention-to-treat principle. If appropriate, multiple imputation methods will be applied (using data from social and medical national registries coupled with health check data), and sensitivity analyses will be performed. Moreover, the potential effect of clustering by the general practitioners will be investigated. The statistical significance level is set at p < 0.05.

ETHICS AND LEGAL ASPECTS

The trial will comply with The Declaration of Helsinki and each participant will provide written informed consent for data to be used for research purposes in agreement with the Danish Health Law. Approval by The Danish Data Protection Agency is obtained (2013-41-2527).

ELIGIBILITY:
Inclusion Criteria:

* Citizens in the municipality of Randers per 01.01.2012
* Randomized for the third group of five to be invited for a preventive health check as part of the health promotion program, Check your health prevention program, conducted in the years 2012 to 2017.
* Having received a preventive health check before November 30 2015.
* Having consented for data to be used scientifically.

Exclusion Criteria:

* Terminal illness as reported by the citizens general practitioner.

Ages: 30 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2201 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | One-year follow up
  Mean cardiorespiratory fitness level and the percentage of participants with very low cardiorespiratory fitness level assessed at the one year follow up will be compared between the two study groups.

SECONDARY OUTCOMES:
Reported physical inactivity prevalence change | Between baseline and the one-year follow up.
  Change in reported physical inactivity prevalence from baseline to one-year follow up will be compared between the two study groups.
Self-rated general health change | From baseline to the one-year follow up.
  Change in self-rated general health from baseline to the one-year follow up will be compared between the two study groups.
Self-rated physical health score change | From baseline to the one-year follow up.
  Change in self-rated physical health scores from baseline to the one-year follow up will be compared between the two study groups.
Self-rated mental health score change | From baseline to the one-year follow up.
  Change in self-rated mental health scores from baseline to the one-year follow up will be compared between the two study groups.

OTHER OUTCOMES:
Stages of Change for physical activity | From baseline to an intermediate two-weeks follow up.
  Stages of Change will be assessed at baseline and two weeks after the health check. Transitions in Stages of Change will be compared between study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Annelli Sandbæk, Professor, Study Chair — Institute of public health, section of general practice, Aarhus University
Locations (1):
- Institute of public health, section of general practice, Aarhus University, Aarhus C, Aarhus County, Denmark

REFERENCES:
- [Background] DISHMAN R, ICKES W, MORGAN W. Self-motivation and adherence to habitual physical-activity. J Appl Soc Psychol. 1980;10(2):115-132. doi: 10.1111/j.1559-1816.1980.tb00697.x.
- [Background] Dalton AR, Soljak M. The nationwide systematic prevention of cardiovascular disease: the UK's health check programme. J Ambul Care Manage. 2012 Jul-Sep;35(3):206-15. doi: 10.1097/JAC.0b013e318240be9d. PMID 22668610
- [Background] Lauritzen T, Jensen MS, Thomsen JL, Christensen B, Engberg M. Health tests and health consultations reduced cardiovascular risk without psychological strain, increased healthcare utilization or increased costs. An overview of the results from a 5-year randomized trial in primary care. The Ebeltoft Health Promotion Project (EHPP). Scand J Public Health. 2008 Aug;36(6):650-61. doi: 10.1177/1403494807090165. PMID 18775821
- [Background] Warburton DE, Nicol CW, Bredin SS. Health benefits of physical activity: the evidence. CMAJ. 2006 Mar 14;174(6):801-9. doi: 10.1503/cmaj.051351. PMID 16534088
- [Background] Textbook of work physiology. Åstrand & Rodahl. 3rd ed. McGraw Hill 1986.
- [Background] Nigg CR. There is more to stages of exercise than just exercise. Exerc Sport Sci Rev. 2005 Jan;33(1):32-5. PMID 15640718
- [Background] Saltin B, Grimby G. Physiological analysis of middle-aged and old former athletes. Comparison with still active athletes of the same ages. Circulation. 1968 Dec;38(6):1104-15. doi: 10.1161/01.cir.38.6.1104. No abstract available. PMID 5721960
- [Background] Ware JE, Kosinski M, Turner-Bowker DM, Gandeck B, eds. User∩s manual for the SF-12v2TM health survey (with a supplement documenting the SF-12 health survey). Lincoln, RI: QualityMetric Incorporated, 2007; 2007.
- [Background] Waters L, Reeves M, Fjeldsoe B, Eakin E. Control group improvements in physical activity intervention trials and possible explanatory factors: a systematic review. J Phys Act Health. 2012 Aug;9(6):884-95. doi: 10.1123/jpah.9.6.884. PMID 22898467
- [Background] Adams G, Gulliford MC, Ukoumunne OC, Eldridge S, Chinn S, Campbell MJ. Patterns of intra-cluster correlation from primary care research to inform study design and analysis. J Clin Epidemiol. 2004 Aug;57(8):785-94. doi: 10.1016/j.jclinepi.2003.12.013. PMID 15485730
- [Background] Sterne JA, White IR, Carlin JB, Spratt M, Royston P, Kenward MG, Wood AM, Carpenter JR. Multiple imputation for missing data in epidemiological and clinical research: potential and pitfalls. BMJ. 2009 Jun 29;338:b2393. doi: 10.1136/bmj.b2393. PMID 19564179
- [Derived] Hoj K, Skriver MV, Hansen AL, Christensen B, Maindal HT, Sandbaek A. Effect of including fitness testing in preventive health checks on cardiorespiratory fitness and motivation: study protocol of a randomized controlled trial. BMC Public Health. 2014 Oct 10;14:1057. doi: 10.1186/1471-2458-14-1057. PMID 25300392
- See also: World Health Organization. Global action plan for the prevention and control of noncommunicable diseases 2013-2020 — http://apps.who.int/iris/bitstream/10665/94384/1/9789241506236_eng.pdf?ua=1.